CLINICAL TRIAL: NCT06319768
Title: Efficacy of Intralesional Injection of Pentoxifylline, Platelet-Rich Plasma, and Combined
Brief Title: Efficacy of Intralesional Injection of Pentoxifylline, Platelet-Rich Plasma, and Combined Pentoxifylline With Platelet-Rich Plasma in Patients With Atrophic Acne Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Mossad Soliman, resident of Dermatology at Kom Ombu Central Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-24-01-04ms
Record Dates: First submitted 2024-02-25; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Atrophic Acne Scar
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- - In group A (PTX group) (n:25): (Active Comparator): Patients will be treated with intralesional PTX (Trentoximal Ampoule 100 mg/5 ml) in a dose of 1mg per lesion at a distance 1cm between two atrophic lesions with a maximum 20 mg per session (with insulin syringe 30Gx8mm). Lesion blanching is the endpoint of injection.
  Interventions: Drug: Pentoxifylline
- - In group B(PRP group) (n:25): (Active Comparator): Patients will be treated with intralesional PRP. PRP will be obtained by the double-spin method, followed by the collection of 10 mL of autologous whole blood into tubes containing trisodium citrate as an anticoagulant. The collected blood will first be centrifuged at 1000 RPM for 10 minutes at room temperature to separate the red blood cells at the bottom of the tube, the buffy coat (containing the white blood cells) in the middle, and the plasma above (soft spin). Then, the upper plasma will be pipetted above the buffy coat to undergo another centrifugation at 1500 RPM for another10 minutes (hard spin) to obtain a platelet pellet in the bottom of the tube (with a platelet count 4-4.5 times higher than that of baseline) and a platelet-poor plasma(PPP) in the upper part. The PPP will be partly removed and partly used to re-suspend the platelets to finally produce 2 mL of PRP.
  Interventions: Drug: platelet rich plasma
- - In group C (combined PTX & PRP) (n:25): (Active Comparator): Patients will be treated with a combination of both intralesional 1mg of PTX per lesion (with a maximum 20mg per session) then 0.1ml of intralesional PRP at the same lesion after 5 minutes.
  Interventions: Drug: combined pentoxifylline and platelet rich plasma

INTERVENTIONS:
Drug: Pentoxifylline — Patients will be treated with intralesional PTX (Trentoximal Ampoule 100 mg/5 ml) in a dose of 1mg per lesion at a distance 1cm between two atrophic lesions with a maximum 20 mg per session (with insulin syringe 30Gx8mm). Lesion blanching is the endpoint of injection
  Arms: - In group A (PTX group) (n:25):
Drug: platelet rich plasma — Patients will be treated with intralesional PRP. PRP will be obtained by the double-spin method, followed by the collection of 10 mL of autologous whole blood into tubes containing trisodium citrate as an anticoagulant. The collected blood will first be centrifuged at 1000 RPM for 10 minutes at room temperature to separate the red blood cells at the bottom of the tube, the buffy coat (containing the white blood cells) in the middle, and the plasma above (soft spin). Then, the upper plasma will be pipetted above the buffy coat to undergo another centrifugation at 1500 RPM for another10 minutes (hard spin) to obtain a platelet pellet in the bottom of the tube (with a platelet count 4-4.5 times higher than that of baseline) and a platelet-poor plasma(PPP) in the upper part. The PPP will be partly removed and partly used to re-suspend the platelets to finally produce 2 mL of PRP
  Arms: - In group B(PRP group) (n:25):
Drug: combined pentoxifylline and platelet rich plasma — Patients will be treated with a combination of both intralesional 1mg of PTX per lesion (with a maximum 20mg per session) then 0.1ml of intralesional PRP at the same lesion after 5 minutes
  Arms: - In group C (combined PTX & PRP) (n:25):

SUMMARY:
Platelet-rich plasma (PRP) is an Acne vulgaris is a common chronic inflammatory skin disorder. It is the eighth most prevalent disease worldwide with a prevalence of 9.4%. Acne scar is one of the most persistent complications of acne, causes marked psychological stress to the patient . The process of acne scar formation can be broadly divided into two stages: increased tissue formation and loss or damage of tissue, corresponding to keloid or hypertrophic scar and atrophic scar, respectively.

The ultimate severity of acne scars is correlated with acne grade and the delay in treatment of active disease. The atrophic scars include three subtypes: icepick or V-shaped, rolling or M-shaped, and boxcar or U-shaped scars. Among atrophic scars, the ice pick type represents 60%-70%; the boxcar type represents 20%-30%; and the rolling type represents 15%-25% (Salameh and Shumaker, 2022). According to the qualitative scarring grading system, a macular acne scar type also exists, which clinically shows erythematous, hyperpigmented, or hypopigmented flat marks.

autologous blood product containing high concentrations of platelets in a small volume of plasma. PRP has been utilized in the treatment of orthopedic, musculoskeletal, and maxillofacial conditions for many years, it has only recently gained popularity in dermatology. PRP contains various growth factors, including platelet-derived growth factor (PDGF), transforming growth factor (TFG), vascular endothelial growth factor (VEGF), and insulin-like growth factor (IGF). These growth factors stimulate tissue remodeling and are associated with enhanced healing through the attraction of macrophages, upregulation of collagen synthesis, and promotion of tissue regeneration. Moreover, platelet-derived growth factor (PDGF) was shown to promote wound healing, angiogenesis, and tissue remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old.
* Both sexes.
* All types of atrophic acne scars

Exclusion Criteria:

* • Pregnant or lactating women.

  * Coagulation disorders or anemia.
  * Skin infections.
  * Patients with hormonal disturbance.
  * Chronic disease e.g: diabetes, renal disease….etc.
  * Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
goodman and baron qualitative grading system of postacne scarring | 6 months
  * The physician's clinical assessment will be performed for all groups by grading the scars before the treatment at baseline, after each treatment session, and 3 months after the last session. Any changes in scar grading will be documented using the Goodman and Baron qualitative acne scarring grading system, with four grades: Grade 1 states the macular scars. Grades 2, 3, and 4 represent mild, moderate, and sever atrophic acne scars, respectively
  * Group B (n: 25): Will receive intralesional injection of PRP.
  * Group C (n: 25): Will receive combined intralesional injection of both PTX & PRP.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Alves R, Grimalt R. Platelet-Rich Plasma and its Use for Cicatricial and Non-Cicatricial Alopecias: A Narrative Review. Dermatol Ther (Heidelb). 2020 Aug;10(4):623-633. doi: 10.1007/s13555-020-00408-5. Epub 2020 Jun 17. PMID 32557337
- [Background] Balazic E, Axler E, Konisky H, Khanna U, Kobets K. Pentoxifylline in dermatology. J Cosmet Dermatol. 2023 Feb;22(2):410-417. doi: 10.1111/jocd.15445. Epub 2022 Oct 31. PMID 36208009
- [Background] Bhargava S, Kroumpouzos G, Varma K, Kumar U. Combination therapy using subcision, needling, and platelet-rich plasma in the management of grade 4 atrophic acne scars: A pilot study. J Cosmet Dermatol. 2019 Aug;18(4):1092-1097. doi: 10.1111/jocd.12935. Epub 2019 Mar 28. PMID 30924301
- [Background] Connolly D, Vu HL, Mariwalla K, Saedi N. Acne Scarring-Pathogenesis, Evaluation, and Treatment Options. J Clin Aesthet Dermatol. 2017 Sep;10(9):12-23. Epub 2017 Sep 1. PMID 29344322